CLINICAL TRIAL: NCT04087577
Title: Effects of Motor Learning After Upper Limb Peripheral Nerve Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 201900433A3
Record Dates: First submitted 2019-08-26; First posted 2019-09-12 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2020-07

CONDITIONS: Peripheral Nerve Injury at Forearm Level (Diagnosis)
Keywords: peripheral nerve injury; motor learning; mirror therapy; physical therapy
MeSH Terms: conditions — Disease; Peripheral Nerve Injuries | interventions — Mirror Movement Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): conventional physical therapy with mirror therapy
  Interventions: Other: conventional physical therapy; Other: mirror therapy
- control group (Active Comparator): conventional physical therapy
  Interventions: Other: conventional physical therapy

INTERVENTIONS:
Other: conventional physical therapy — includes electrical stimulation for denervated muscles, and soft tissue massage, joint range of motion exercises to maintain the flexibility of the affected joint, muscle or connected tissues, sensory relearning
Other: mirror therapy — mirror therapy
  Arms: experimental group

SUMMARY:
The outcome of peripheral nerve injury is related to age, level of injury, the injured nerve, the severity of injury, and the timing and the type of surgery interventions. In addition, high-level peripheral nerve injury would not full recovery, and the prognosis is determined by the nerve regeneration.

Conventional physical therapy includes electrical stimulation for denervated muscles, and soft tissue massage, joint range of motion exercises to maintain the flexibility of the affected joint, muscle or connected tissues. However, the nerve regeneration takes several months in high-level median, ulnar or radial nerve injury. Prolonged median or ulnar nerves injury may interfere intrinsic muscular function, and radial nerve injury causes drop hand. Earlier nerve regeneration or motor training is essential for the patients to return to normal life and increase their quality of life

DETAILED DESCRIPTION:
The outcome of peripheral nerve injury is related to age, level of injury, the injured nerve, the severity of injury, and the timing and the type of surgery interventions. In addition, high-level peripheral nerve injury would not full recovery, and the prognosis is determined by the nerve regeneration.

Conventional physical therapy includes electrical stimulation for denervated muscles, and soft tissue massage, joint range of motion exercises to maintain the flexibility of the affected joint, muscle or connected tissues. However, the nerve regeneration takes several months in high-level median, ulnar or radial nerve injury. Prolonged median or ulnar nerves injury may interfere intrinsic muscular function, and radial nerve injury causes drop hand. Earlier nerve regeneration or motor training is essential for the patients to return to normal life and increase their quality of life. This research aims to explore the effects of mirror therapy for peripheral nerve injury. We will enroll 60 patients who suffer from median, ulnar or radial nerve injury at the level of elbow or proximal forearm. The subjects will be randomized into the mirror-therapy group or the control group. Each group will receive conventional physical therapy (i.e., electrical stimulation, joint range of motion exercise, muscle strengthening training, sensory reeducation training). The mirror-therapy group would be supplemented by motor learning by mirror therapy. The measurements include joint range of motion, pain status, sensibility, grip strength, pinch strength, hand function test and the Disabilities of the Arm, Shoulder and Hand (DASH). Demographic information will be collected and analyzed by the independent t-tests. The outcome variables taken during the three and six months after the interventions would be included. One-way ANOVA are used to compare the difference between measurements. This study may offer an evidence based results to explore the effects of mirror therapy for peripheral nerve regeneration and motor learning.

ELIGIBILITY:
Inclusion Criteria:

* Willing to sign the inform consent
* Sufficiently communicate in the Chinese language
* Be able to follow instructions
* Newly median, ulnar, or radial nerve repair at forearm level in recent 3 weeks

Exclusion Criteria:

* Pregnant or breast-feeding woman
* Central nervous disease
* A history of nerve entrapment syndrome in recent 1 year
* Patients with a history of latent neuropathy, such as diabetes, dialysis, and tumor
* Unable to communicate or comprehend the questionnaires

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-12-19 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
change from baseline in Semmes-Weinstei monofilaments (SWM) at 3 and 6 months | baseline, 3 months, 6 months
  force in grams
change from baseline in two-point discrimination (2PD) at 3 and 6 months | baseline, 3 months, 6 months
  S0-4, higher score indicates better outcome
change from baseline in grip power at 3 and 6 months | baseline, 3 months, 6 months
  grip power in kilograms

SECONDARY OUTCOMES:
change from baseline in upper-extremity functional outcomes at 3 and 6 months | baseline, 3 months, 6 months
  The Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire ranges from 0-100. Lower score indicates better outcomes.
Minnesota rate of manipulation tests | baseline, 3 months and 6 months
  Manipulation tests in seconds
Purdue Pegboard Test | baseline, 3 months and 6 months
  Manipulation tests in seconds
functional MRI activation | 3 months
  movement and sensory tests to calcuate z-score by software

CONTACTS AND LOCATIONS:
Overall Officials: Yueh-Hsia Chen, Master, Principal Investigator — Chang Gung Memorial Hospital
Locations (2):
- Taiwan (2):
  - Department of Plastic and Reconstructive Surgery Rehabilitation Center, Chung Gung Memorial Hospital, Taoyuan District
  - Chang Gung Memorial Hospital, Taoyuan District